CLINICAL TRIAL: NCT04703426
Title: Copy of A Phase II Trial of Pembrolizumab (Anti PD-1) Therapy Combined With Sargramostim (GM-CSF) in Unresectable or Metastatic Melanoma
Brief Title: Sargramostim (GM-CSF) + PD-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Partner Therapeutics (PTx) (Unknown)
Responsible Party: Principal Investigator, Elizabeth Buchbinder, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-370
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Unresectable Melanoma; Metastatic Melanoma; Stage III Melanoma; Stage IV Melanoma
Keywords: Unresectable Melanoma; Metastatic Melanoma; Stage III Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sargramostim (GM-CSF) + Pembrolizumab (anti-PD-1) (Experimental): Participants will receive 12 weeks of sargramostim (GM-CSF) and pembrolizumab (anti-PD-1). Participants may be pre-medicated with drugs to reduce the chance of having a sensitivity reaction to the study treatment of pembrolizumab (anti-PD-1) and sargramostim (GM-CSF).
  Study cycles are 21 days in length:
  * Pembrolizumab (anti-PD-1) will be given by intravenous infusion once on day 1 of every 21 day cycle
  * Sargramostim (GM-CSF) will be self-administered by participants via a subcutaneous (below the skin) injection daily for days 1 - 14 of each 21- day cycle.
  Participants will be assessed at 12 weeks for disease response/progression and further study treatment.
  Interventions: Drug: Sargramostim (GM-CSF); Drug: Pembrolizumab (anti-PD-1)

INTERVENTIONS:
Drug: Sargramostim (GM-CSF) — Drug that binds to the protein PD-1 to help immune cells kill cancer cells better, it is given as an intravenous injection through a vein.
  Other Names: Leukine
Drug: Pembrolizumab (anti-PD-1) — Drug that stimulates blood cells that may help support the immune system during cancer treatment, given as intravenous infusion
  Other Names: Keytruda

SUMMARY:
This research study is testing the combination of two drugs, sargramostim and pembrolizumab. The study is designed to see if the combination of these study drugs would improve the control of unresectable or metastatic melanoma cancer when compared to use of these drugs alone.

The names of the study drugs involved in this study are:

* Pembrolizumab
* Sargramostim (GM-CSF)

DETAILED DESCRIPTION:
This is an open-label phase II study looking at safety and efficacy of the combination of pembrolizumab (PD-1 inhibition and sargramostim (GMCSF) in people with unresectable stage III or IV melanoma who may have received prior immunotherapy in the metastatic setting.

The U.S. Food and Drug Administration (FDA) has not approved sargramostim as a treatment option for people with stage III or IV melanoma The U.S. Food and Drug Administration (FDA) has approved pembrolizumab as a treatment option for people with stage III or IV melanoma who have received prior immunotherapy in the metastatic setting.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive the study drug(s) for as long as they do not have serious side effects and their disease does not get worse and will be followed for safety 30 days after the last dose of study drug(s). Participants may also be followed for long term follow-up every 12 weeks from the last dose of study drug(s).

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of metastatic or unresectable stage III or IV cutaneous melanoma
* Prior treatment with immunotherapy
* Age ≥ 18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Measurable disease (by CT, PET/CT or MRI)
* The effects of GMCSF and PD-1 inhibition on the developing human fetus are unknown.

For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 7 months after completion of study drug administration.

* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases must have documented stability over a four week interval and not be requiring active treatment for these. Prior radiation, surgery and stereotactic radiosurgery are allowed but must be completed four weeks prior to initiating therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pembrolizumab or sargramostim.
* Need for systemic steroids at the time of enrollment. Physiologic replacement at a dose of less than 10mg daily prednisone equivalent is allowed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants who are considered Women of Child-Bearing Potential (WOCBP) must have a negative serum pregnancy test in order to be eligible. Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Pembrolizumab, breastfeeding should be discontinued if the mother is treated with Pembrolizumab. These potential risks may also apply to other agents used in this study.
* Known active HIV, Hepatitis B or Hepatitis C patients. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for an immunologic effect with the therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Autoimmune disease that requires treatment at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 12 weeks
  The primary study endpoint is response rate per RECIST criteria.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 12 weeks
  Number and proportion of adverse events, graded as defined by CTCAE version 5.0
Overall Survival Rate | 12 weeks
  Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) will be used.
Progression Free Survival Rate | 12 weeks
  Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) will be used.
Overall Response Rate (ORR)-irRC | 12 weeks
  To evaluate the overall response rate in advanced melanoma to combination anti- PD-1 therapy and sargramostim by irRC criteria.
CD4+ ICOS T cell changes | 12 weeks
  Evaluate changes in CD4+ ICOS T cells from biopsies (pre-treatment, on-treatment, post-treatment) and correlate using Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Buchbinder, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu